CLINICAL TRIAL: NCT03520738
Title: Arterial Calcifications: Role of Tissue-nonspecific Alkaline Phosphatase in Phosphate and Pyrophosphate Homeostasis. PIPAL Study.
Brief Title: Tissue-nonspecific Alkaline Phosphatase in Phosphate and Pyrophosphate Homeostasis.
Acronym: PIPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-AOIP-01
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronic Kidney Disease (Other): Blood and urinary samples on the following patients:
  10 Stage 1 and 2 CKD patients 10 patients 6 weeks after graft 10 patients on maintenance dialysis.
  Interventions: Other: Blood samples; Other: Urinary samples
- Pseudoxanthoma elasticum (PXE) (Other): Blood and urinary samples on the following patients:
  10 patients with pseudoxanthoma elasticum (PXE) with low PPi levels and vascular calcifications and patients with hypophosphatasia (HPP) with high PPi levels and bone decalcification.
  Interventions: Other: Blood samples; Other: Urinary samples
- Hypophosphatasia (HPP) (Other): Blood and urinary samples on the following patients:
  4 patients with hypophosphatasia (HPP) with high PPi levels and bone decalcification.
  Interventions: Other: Blood samples; Other: Urinary samples

INTERVENTIONS:
Other: Blood samples — Blood samples on an empty stomach
Other: Urinary samples — first urinary in the morning

SUMMARY:
Vascular calcification is a common finding in chronic kidney disease and increases arterial stiffness leading to augmented cardiovascular morbidity. The calcification process is thoroughly regulated by pro and anticalcifying agents. The investigators hypothesize that imbalance in these compounds could depend on alkaline phosphatase activity. Therefore, the investigators will measure ALP activity, calcifications score, arterial stiffness and perform a bio-collection in monogenic rare diseases characterized by various levels of anticalcifying agents and in diverse CKD stages characterized by various levels of procalcifying compounds.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) describes the gradual loss of kidney function from stage 1 (normal renal function) to stage 5 requiring maintenance dialysis or kidney transplantation (KT). Vascular calcification in CKD is a common finding and increases arterial stiffness leading to increased cardiovascular morbidity. The calcification process is the same for bones and arteries and is thoroughly regulated by pro and anticalcifying agents. Actually, inorganic phosphates (Pi) accelerate the calcification process and their levels are found increased in advanced CKD stage. In contrast, inorganic pyrophosphates (PPi) are potent anti-calcifying compounds resulting from the hydrolysis of extracellular ATP, but their role in CKD remains elusive. Tissue-nonspecific alkaline phosphatases (TNAP) convert PPi into Pi in calcification sites leading to hydroxyapatite deposition. The metabolism of PPi depends on diverse compounds, which are included in our bio-collection (Favre, Int J Mol Sci, 2017). The activity of plasma Alkaline Phosphatase (ALP) reflects the tissue production of TNAP. ALP activity is correlated to cardiovascular events in CKD patients. Preliminary results from our group show a stable plasma level of the PPi/Pi ratio independently from the glomerular filtration rate.

The investigators hypothesize that PPi/Pi imbalance could depend on ALP activity and could be a key determinant of vascular calcifications and arterial stiffness.

Therefore, the investigators will measure ALP activity, calcifications score, arterial stiffness and perform a bio-collection in monogenic rare diseases and in various CKD stages including hyperphosphatemic patients on maintenance hemodialysis.

Stage 1 and 2 CKD patients will be considered as a reference group because Pi levels and PPi levels are usually normal and calcification level is low. These patients will be compared to CKD patients with various Pi levels : low Pi levels in KT recipients 6 weeks after graft and high Pi levels in patients on maintenance dialysis. These patients (CKD 1 and 2) will be compared to patients with various PPi levels: patients with pseudoxanthoma elasticum (PXE) with low PPi levels and vascular calcifications and patients with hypophosphatasia (HPP) with high PPi levels and bone decalcification. PXE and HPP are rare monogenic disorder resulting from mutation in ABCC6 and the gene encoding TNAP respectively.

ELIGIBILITY:
Inclusion Criteria:

* patient with Chronic kidney disease (stage 1 or 2, 6 weeks after graft or patients on maintenance dialysis) or patient with pseudoxanthoma elasticum or patient with hypophosphatasia
* informed consent signed

Exclusion Criteria:

* cancer
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
ALP activity (alkaline phosphatase activity) | at time = day 0 (inclusion)
  ALP activity will be plotted against the PPi/Pi ratio in CKD patients with various Pi levels; a regression curve will be used to measure the correlation between these two factors

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FAVRE, MD, Principal Investigator — Nephrology Department, Nice University Hospital
Locations (4):
- France (4):
  - CHU d'Angers - Service de Dermatologie, Angers
  - Service de Médecine Vacsulaire - CHU d'ANGERS, Angers
  - CHU de Nice, Nice
  - Service de Rhumatologie - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No